CLINICAL TRIAL: NCT04669886
Title: Serum Endotoxin Assay to Predict the Development of Postoperative Infectious Complications and Systemic Inflammatory Response Following Percutaneous Nephrolithotomy.
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hemendra Shah, Associate Professor of clinical Urology, University of Miami
Other Study IDs: 20200234
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Nephrolithiasis; Urosepsis
Keywords: endotoxin; fever; infectious complications; endourology; percutaneous nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endotoxin study group: Patients scheduled for Percutaneous Nephrolithotomy (PCNL) as surgical treatment for their kidney stones will be evaluated for postoperative endotoxin levels as a risk marker for sepsis.

SUMMARY:
The aim of the study is to establish an infectious risk stratification system based on pre-and post-operative blood endotoxin profile.

ELIGIBILITY:
Inclusion Criteria:

* Adults that is able to consent (≥ 18 years of age)
* Scheduled to undergo PCNL at Uhealth tower and Jackson Memorial Hospitals
* not currently immunosuppressed [White blood count (WBC) >= 2, not on immunosuppressive medications]

Exclusion Criteria:

* unable to consent and < 18 years of age
* currently immunosuppressed (WBC < 2, not on immunosuppressive medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for PCNL as surgical treatment for their kidney stones at Jackson and the University of Miami Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants at each endotoxin activity level after surgery. | Day 1 (within 30 minutes postoperative)
  The endotoxin activity level assessed from blood samples will be categorized as low (<0.40), intermediate (0.40-0.59) or high (≥0.60) endotoxin activity level. Analysis will be done via Endotoxin Activity Assay (EAA).
Corelation of endotoxin activity level with post-operative infectious complication | up to 24 hours
  infectious complications include fever, and signs and symptoms of systemic inflammatory response syndrome as evaluated by treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Hemendra N Shah, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No